CLINICAL TRIAL: NCT04632446
Title: Upgrade Program Implementation at Colorrectal Surgery and Complications: Early Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Other Study IDs: IMIB-2020-UPCS
Record Dates: First submitted 2020-10-28; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Early diagnosis — Early diagnosis. Upgrade program implementation.

SUMMARY:
The anastomotic leak (AL) is a very serious complication in colorectal surgery not only because of its severity but its frequency. Other facet for study, besides the risk factor and prevention, is the AL early diagnostic, due to minimize the clinical consequences and severity; and avoid the failure-to-recue. Several studies analyze the Creactive protein (CRP) and Procalcitonine (PCT) usefulness in AL predictor before the clinical signs appear.

At a prospective observational study carry on our center, it concluded that CRP at 3rd day after surgery over 15mg/dl was a very important AL predictor, even before the clinical changes appear. The aim of this study is minimize the severity complications and the mortality due to AL appears. The aim of this study is minimize the severity complications and the mortality due to AL by means of introduces an upgrade program in which a CT scan will be conduct in all the patients with high CRP levels at 3rd, 4th or 5th postoperative day, with the goal to know the AL early and make all the therapeutic step to minimize the consequences.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients undergoing elective colorectal surgery due to neoplastic or non-neoplastic etiology.
* Patients with an anastomosis performed in the surgical act.
* Signed informed consent.

Exclusion Criteria:

* Patients who require transfer to another center.
* Patients with fatal evolution: those who require urgent reoperation for an inarverted perforation, early leakage of anastomosis or death before the third postoperative day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent elective colorectal surgery consecutively will be included, in which an anastomosis have been performed (neoplastic and non-neoplastic pathology
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Severity of morbidity | 1 year
  Number of reoperations, readmissions for infections associated or other medical complications, terminal stomata
Severity of mortality | 1 year
  Number of related exits

SECONDARY OUTCOMES:
- Compare hospital stay and ICU stay of patients undergoing elective colorectal surgery before and after the improvement program. | 1 year
- Evaluate the difference in the incidence of anastomosis leak after the implementation of the improvement program | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Graciela Valero-Navarro, MD, Principal Investigator — - Hospital Morales Meseguer
Locations (1):
- - Hospital Morales Meseguer, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baeza-Murcia M, Valero-Navarro G, Pellicer-Franco E, Soria-Aledo V, Mengual-Ballester M, Garcia-Marin JA, Betoret-Benavente L, Aguayo-Albasini JL. Early diagnosis of anastomotic leakage in colorectal surgery: prospective observational study of the utility of inflammatory markers and determination of pathological levels. Updates Surg. 2021 Dec;73(6):2103-2111. doi: 10.1007/s13304-021-01082-8. Epub 2021 May 20. PMID 34018141